CLINICAL TRIAL: NCT02052206
Title: Reconstruction of Complex Proximal Humeral Fractures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Lazaros Vlachopoulos, MD, MD, Balgrist University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BalgristUH_CARD_03
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis of the Shoulder; Complexe Proximal Humeral Fractures
Keywords: osteoarthritis; complexe proximal humeral fracture; shoulder; shoulder replacement; accuracy; computer-assisted; 3D
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Computer-assisted 3D planning (Experimental): Realization of the fracture reconstruction according to the computer-assisted 3D preoperative plan
  Interventions: Procedure: Shoulder replacement surgery

INTERVENTIONS:
Procedure: Shoulder replacement surgery

SUMMARY:
The purpose of this study is to evaluate the accuracy of shoulder replacement surgery in realization a computer assisted 3D planning compared to conventional 2D planning.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis or complexe proximal humeral fracture and indication for shoulder arthroplasty
* patients > 18years

Exclusion Criteria:

* contraindication for computertomography
* pregnancy
* previous fracture or shoulder replacement of the contralateral side in case of a complexe proximal humeral fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Quantitative analysis of the accuracy of an automatic algorithm for the reconstruction of proximal humeral fractures | 6 weeks
  Accuracy of the reconstruction of complex proximal humeral fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Lazaros Vlachopoulos, MD, Study Chair — Balgrist University Hospital
Locations (1):
- University Hospital Balgrist, Zurich, Switzerland

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196